CLINICAL TRIAL: NCT03402165
Title: Impact of Serum Alpha-fetoprotein Levels on the Response to Direct Antiviral Therapy in Egyptian Patients With Chronic Hepatitis C
Brief Title: Serum Alpha-fetoprotein Levels and Response to Direct Antiviral Therapy in Patients With Chronic Hepatitis C
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alfafetoprotein
Record Dates: First submitted 2018-01-09; First posted 2018-01-18 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Alfafetoprotein (Experimental): Sofosbuvir and Ledipasvir or sofosbuvir and daklatasuvir
  Interventions: Drug: Sofosbuvir and Ledipasvir or sofosbuvir and daklatasuvir
- Mild elevation of alfafetoprotein (Experimental): Sofosbuvir and Ledipasvir or sofosbuvir and daklatasuvir
  Interventions: Drug: Sofosbuvir and Ledipasvir or sofosbuvir and daklatasuvir
- High elevation of alfafetoprotein (Experimental): Sofosbuvir and Ledipasvir or sofosbuvir and daklatasuvir
  Interventions: Drug: Sofosbuvir and Ledipasvir or sofosbuvir and daklatasuvir

INTERVENTIONS:
Drug: Sofosbuvir and Ledipasvir or sofosbuvir and daklatasuvir — Response to DAAD's and developing HCC
  Other Names: Sofaldy, Harvony

SUMMARY:
Alpha-fetoprotein Levels on the Response to direct Antiviral Therapy in Patients with Chronic Hepatitis C

DETAILED DESCRIPTION:
Impact of Serum Alpha-fetoprotein Levels on the Response to direct Antiviral Therapy in Egyptian Patients with Chronic Hepatitis C

ELIGIBILITY:
Inclusion Criteria:

* HCV patients who will undergo treatment by direct acting antiviral agents.

Exclusion Criteria:

* Patients with decompensated liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with sustained virologic response | 6 months
  The total number of patients with SVR in each group

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Badawi, MD, Principal Investigator — Tanta University; Mohamed Alboraie, MD, Study Director — Al-Azhar University; Sherief Abd-Elsalam, MD, Study Director — Tanta University; Mohamed el kassas, MD, Study Director — Helwan University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided